CLINICAL TRIAL: NCT00882414
Title: A Multi-centre, Randomized, Controlled, Single-blinded, Phase II Study to Investigate the Safety and Efficacy of Intravenous Infusions of FERINJECT® Versus Placebo in Patients With Thrombocytosis Secondary to Iron Deficiency and Chronic Inflammatory Bowel Disease
Brief Title: Ferinject® in Patient With Thrombocytosis Secondary to Inflammatory Bowel Disease (IBD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Main objective of study was met. Further recruitment was difficult.
Sponsor: Vifor Pharma (Industry)
Responsible Party: Lise Riopel PhD/Clinical Indication Leader, Vifor (International) Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THROMBOVIT
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Thrombocytosis; Iron-Deficiency Anemia
Keywords: ferric carboxymaltose; platelet; thrombocyte; ferritin; hemoglobin; transferrin
MeSH Terms: conditions — Thrombocytosis; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- ThromboVIT Placebo (Placebo Comparator): Patients will receive 1 placebo infusion of 100ml 0.9% sodium chloride every 7 days for a total of 3 infusions.
  Interventions: Drug: Placebo
- ThromboVIT 1000 (Experimental): ThromboVIT 1000: Patients will receive 1 infusion of 500mg Ferinject® diluted in 100ml 0.9% sodium chloride every 7 days for a total of 2 infusions (1000 mg) followed by 1 placebo infusion of 100ml 0.9% sodium chloride.
  Interventions: Drug: FERINJECT® (Ferric carboxymaltose)
- ThromboVIT 1500 (Experimental): Patients will receive 1 infusion of 500mg Ferinject® diluted in 100ml 0.9% sodium chloride every 7 days for a total of 3 infusions (1500 mg).
  Interventions: Drug: FERINJECT® (Ferric carboxymaltose)
- ThromboVIT 500 (Experimental): ThromboVIT 500: Patients will receive 1 infusion of 500mg Ferinject® diluted in 100ml 0.9% sodium chloride (500 mg) followed by 2 placebo infusions of 100ml 0.9% sodium chloride every 7 days.
  Interventions: Drug: FERINJECT® (Ferric carboxymaltose)

INTERVENTIONS:
Drug: FERINJECT® (Ferric carboxymaltose) — FERINJECT® will be administered i.v. into a peripheral vein in the arm. 500 mg FERINJECT® will be diluted to a total volume of 100mL in 0.9% saline for infusion and administered over 15 minutes duration.
  Other Names: FERINJECT®
  Arms: ThromboVIT 1000; ThromboVIT 1500; ThromboVIT 500
Drug: Placebo — Placebo will be administered i.v. into a peripheral vein in the arm. A total volume of 100mL 0.9% saline will be administered over 15 minutes duration.
  Other Names: NaCl 0.9%; saline
  Arms: ThromboVIT Placebo

SUMMARY:
The aim of this study is to show the benefits for patients, with a high platelet count, iron deficiency and IBD, receiving intravenous iron therapy.

DETAILED DESCRIPTION:
For the first time a platelet abnormality in IBD was reported in 1968, with a description of an increased platelet count in patients having an exacerbation of clinical activity 1. Since then it has been established that thrombocytosis and platelet activation are common features in IBD2. Both features are strongly connected to thromboembolic events, which are a major cause of patient morbidity and mortality 3. In vitro studies have so far shown that spontaneous platelet aggregation is present in more than 30% of IBD patients compared to none of the controls and besides independent of disease severity 4.

Unfortunately the mechanisms behind the abnormal megakaryopoiesis are not completely understood. Nevertheless platelets can store and produce a large amount of inflammatory mediators and are activated by multiple proinflammatory substances. Therefore, platelets are regarded as a major target in the therapy of inflammatory bowel diseases 5. An increase in systemic cytokine levels such as IL-6 or IL-11 may contribute to enhanced platelet production. Also intestinal bleeding and iron deficiency, which are major symptoms of IBD, may have stimulatory effects on megakaryopoiesis 6.

Previously, we observed a normalization of elevated platelet counts in IBD patients with iron deficiency anemia (IDA) upon treatment with intravenous iron sucrose 7. We therefore believe that iron deficiency is causatively involved in the pathogenesis of thrombocytosis in IBD and intend to investigate the effect of intravenous iron therapy on platelet levels and platelet activation markers in patients with IBD and iron deficiency.

Vifor (International) Inc. has developed a new formulation of parenteral iron, FERINJECT® (5% w/v iron carboxymaltose in a solution of water for injection). Based on preclinical toxicity data and clinical experience, FERINJECT® does not cause anaphylactic reactions or liver toxicity. Based on human pharmacokinetic data, the estimated terminal half-life of FERINJECT® is 16 hours. The analysis of a FERINJECT® positron emission tomography (PET) study in six patients each receiving a single dose of 100mg iron as FERINJECT® demonstrated that, during the initial distribution phase, a major proportion of the dose was distributed to the bone marrow . Red cell utilization of iron was found to be high. After 24 days, patients with IDA showed a red cell utilization of 91% to 99%. Various studies demonstrated that FERINJECT® could be safely administered at doses of up to 1000mg, which is a significant advantage of FERINJECT® over iron sucrose.

A multiple-dose phase I/II study in patients with IBD investigating the safety, efficacy, and kinetics of repeated doses of FERINJECT® has been completed. Patients who were treated at our unit (Medical University of Vienna) were also analyzed regarding the effect of VIT45 on platelet counts. Similar to our experience with iron sucrose, we observed a significant drop in thrombocytosis within 8 weeks pointing again to the direct effect of iron on regulating megakaryopoiesis in vivo8.

This study tries to show the benefits for patients, with a high platelet count, iron deficiency and IBD, receiving intravenous iron therapy.

As with all iron preparations, overdosing with respect to the total amount should be avoided. The maximum infused weekly dose of FERINJECT® will be 500 mg. Based on animal toxicity data and patient experience, FERINJECT® does not cause anaphylactic reactions or liver toxicity at the doses intended for use in this study. However, due to the relatively large doses of iron being administered, patients will be monitored carefully throughout the study for symptoms of iron overload.

Potential benefits to the patients include a decrease of the platelet counts, besides a increase in hemoglobin levels and normalization of iron stores.

Primary Objective:

To evaluate the efficacy of FERINJECT® in reducing elevated platelet counts

Secondary Objectives:

To evaluate the effect of FERINJECT® on coagulation and platelet activation parameters To evaluate the efficacy of FERINJECT® in normalizing iron deficiency To evaluate the change of quality in life and disease activity To evaluate the safety of FERINJECT®

ELIGIBILITY:
Inclusion Criteria:

* Male or female, inpatient or outpatient, aged at least 18 years and not more than 60 years.
* Have a platelet count >450G/l
* Transferrin saturation (TfS) <20% or ferritin < 100µg/l
* Previously diagnosed inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Females of child-bearing potential must have a negative urine pregnancy test at screening and be practicing a highly effective method of birth control during the study and for up to 1 month after the last dose of the study medication. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner. Non-childbearing potential includes being surgically sterilized at least 6 months prior to the study or postmenopausal, defined as amenorrhoea for at least 12 months.
* Demonstrate the ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to undergo the required assessments.

Exclusion Criteria:

* CDAI >220, CAI>6
* Significant anemia (hemoglobin <10.5 g/dl), or anaemia not caused by iron deficiency (e.g. anaemia due to cancer or infection)
* Blood transfusions or iron therapy during the previous 4 weeks, or erythropoietin treatment within the 8 weeks prior to enrollment.
* Concomitant therapy with prednisolone above 20mg/d, 6-mercaptopurine, infliximab or azathioprine must have been initiated at least 4 months prior to study and the dose must be stable for at least 8 weeks. Other drugs with known effects on megakaryopoiesis (e.g. interferon-alpha).
* Severe concomitant disease or need for surgery within 8 weeks
* Hemochromatosis or other iron-storage disorders (e.g. thalassemia, siderosis, lead poisoning anaemia, porphyria cutanea tarda)
* Treatment with an investigational drug within the 30 days prior to enrollment
* Active severe infection or malignancy other than carcinoma in situ of the cervix and non-melanoma skin cancer.
* Bone Marrow Disease (MDS, thalassemia, etc)
* Active or chronic liver or kidney disease. Serum albumin <25 g/L or serum creatinine >20 mg/L
* Significant cardiovascular disease, including myocardial infarction within 12 months prior to study inclusion, congestive heart failure NYHA (New York Heart Association) grade III or IV, or poorly controlled hypertension according to the judgment of the investigator. Known hypersensitivity to FERINJECT®
* Positive for HIV 1/HIV 2 antibodies (anti HIV) (HIV: human immunodeficiency virus).
* Positive for hepatitis B surface-antigen (HBsAg), hepatitis C virus antibody (anti HCV) and evidence for active hepatitis, i.e., abnormal liver function test (LFT) results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of FERINJECT® in reducing elevated platelet counts | 6 weeks post baseline
  The primary efficacy endpoint is a decrease of the platelet counts >25% after 6 weeks.

SECONDARY OUTCOMES:
Normalization of platelet levels | 6 weeks post baseline
  Normalization of platelet levels
Change in platelet activation markers (p-selectin, sCD40L), thrombopoietin and reticulated thrombocytes | 6 weeks post baseline
  Change in platelet activation markers (p-selectin, sCD40L), thrombopoietin and reticulated thrombocytes
Change in coagulation parameters (PTT, PT, factors of the intrinsic coagulation pathway) | 6 weeks post baseline
  Change in coagulation parameters (PTT, PT, factors of the intrinsic coagulation pathway)
Change in iron parameters (ferritin, hemoglobin, transferrin, transferrin saturation, soluble transferrin-receptor, hepcidin) | 6 weeks post baseline
  Change in iron parameters (ferritin, hemoglobin, transferrin, transferrin saturation, soluble transferrin-receptor, hepcidin)
Change in quality of life (IBDQ, SF-36, FACT-An or similar) and disease activity | 6 weeks post baseline
  Change in quality of life (IBDQ, SF-36, FACT-An or similar) and disease activity (CDAI, CAI=Clinical activity scores (Rachmilewitz) without endoscopy)
Change in C-reactive protein, ESR, IL-3, IL-6 and IL-11 and calprotectin. | 6 weeks post baseline
  Change in C-reactive protein, ESR, IL-3, IL-6 and IL-11 and calprotectin.
Adverse Events | 6 weeks post baseline
  Adverse Events (AE): type, nature, incidence and outcome.
Vital signs | 6 weeks post baseline
  Vital signs (axillary temperature, blood pressure and heart rate).
Physical examinations | 6 weeks post baseline
  Physical examinations
Clinical laboratory panels | 6 weeks post baseline
  Clinical laboratory panels (haematology/coagulation, clinical chemistry/inflammation, urinalysis).
Discontinuation of treatment due to AEs | 6 weeks post baseline
  • Discontinuation of treatment due to AEs
Pregnancy test | Visit 4
  Pregnancy test
CDAI/CAI | 6 weeks post baseline
  CDAI/CAI

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gasche, MD, Principal Investigator — Allgemeines KrankenHaus, Vienna, Austria
Locations (1):
- Univ. clinic for Internal Medicine, Vienna, Austria